CLINICAL TRIAL: NCT04092946
Title: Home-based Digital Program for Musculoskeletal Disorders: a Large-scale, Multi-disorder, Prospective, Single-arm, Interventional Study
Brief Title: Digital Home-based Rehabilitation for Musculoskeletal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sword Health, SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SH-SA-MSK-US
Record Dates: First submitted 2019-09-06; First posted 2019-09-17 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Musculoskeletal Diseases
Keywords: Home-based rehabilitation; Biofeedback; Telerehabilitation
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: Single-arm, prospective, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with musculoskeletal disorders (Experimental): Tailored digital programs for individuals working for organizations that enter into a commercial agreement with SWORD Health, which acts as a service provider.
  Interventions: Device: Digital intervention

INTERVENTIONS:
Device: Digital intervention — Individuals included will be offered a program based on three pillars: education, cognitive-behavioural therapy (CBT) and therapeutic exercise.
  The therapeutic exercise component will be delivered in the form of exercise sessions to be performed independently by the individual at home using SWORD Phoenix. These programs will have a duration of between 8 and 12 weeks, according to the condition, following pre-defined protocols. These protocols can be adapted to the needs, performance and progress of each individual by their assigned physical therapist. Individuals will be asked to perform at least 3 exercise sessions per week, in different days, but will not be excluded in case of lower adherence.
  In addition to the exercises, the individuals will also have access to educational articles written by the clinical team, as well as to a CBT program delivered through a combination of written articles and pre-recorded audio sessions.

SUMMARY:
The purpose of this study is to assess the acceptance, engagement and outcomes of a digital care program for acute and chronic musculoskeletal conditions affecting the shoulder, elbow, hip, knee, ankle and spine.

DETAILED DESCRIPTION:
SWORD Health has developed a novel digital biofeedback system for home-based physical rehabilitation - SWORD Phoenix- which is an FDA-listed class I medical device. The company has previously conducted two pilot studies (NCT03047252; NCT03045549) comparing a digital rehabilitation program using this device against conventional face-to-face physical therapy. These studies have proven the feasibility, safety and effectiveness of this medical device on rehabilitation after total knee and hip arthroplasty.

SWORD Health is now seeking additional validation of its digital programs on acute and chronic MSK conditions, to assess the acceptance, engagement and outcomes of these clinical programs. This study will also unveil disease-specific human motion patterns that may be used to inform the development of new diagnostic and treatment tools.

Data to be collected on every individual undergoing our programs includes:

1. data that is sourced from the subject through online assessment forms
2. data that is sourced from the subject, collected by the physical therapist managing that subject (i.e. suggestions for improvement);
3. data that is generated by the physical therapist through interaction with the web-based Portal (i.e. session composition in terms of exercises, sets, repetitions, usage or not of external resistance)
4. data generated by the patient through interaction with the mobile app (i.e. pain and fatigue levels, satisfaction)
5. data that is generated automatically by the medical device (i.e. range of motion, compliance)

Collection and objective analysis of the collected data will allow:

1. Monitoring of user needs, engagement and satisfaction to guide further improvements;
2. Analysis of the effectiveness of these digital care programs;
3. Correlation of results with patient's demographic and clinical profiles;
4. Compilation of patient cohorts to increase and disseminate knowledge on each disorder, its progression and response to physical therapy programs;
5. Explore the cost-efficiency of these digital programs
6. Development of novel intelligent tools to assist therapists with patient management.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Suffering from acute (<12 weeks) or chronic (>12 weeks) pain in the neck, low back, shoulder, elbow, hip, knee, ankle or wrist;
* Able to understand study procedures and willing to provide informed consent

Exclusion Criteria:

* Cardiac or respiratory condition incompatible with at least 20 minutes of light to moderate exercise
* Cancer diagnosis or receiving treatment for cancer
* Unexplained weight loss in the last 6 months
* Significant trauma in the area of pain in the last 3 months
* Rapidly progressive loss of strength and/or numbness in the arms/legs in the last 2 weeks
* Unexplained change in bowel or urinary function in the last 2 weeks
* Other known health condition limiting participation in an exercise program involving at least 20 minutes of light to moderate exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48774 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
Neck, lower spine, shoulder, elbow, ankle, hip and knee range of motion | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through Neck, lower spine, shoulder, elbow, ankle, hip and knee range of motion (ROM) (flexion/extension/abduction/rotation), in degrees, as directly retrieved from the angle measurement tool integrated within the medical device.
Neck Disability Index | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the Neck Disability Index.
  The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Oswestry Disability Index | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the Oswestry Disability Index (ODI). \ The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Short version of the Disabilities of the Arm, Shoulder and Hand questionnaire | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the short version of the Disabilities of the Arm, Shoulder and Hand questionnaire (QuickDASH).
  Scoring Formula = ([(sum of n responses)/n] -1)x(25).
Foot and Ankle Ability Measure | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time, measured through the Foot and Ankle Ability Measure (FAAM).
  FAAM is a self-report measure that assesses physical function of individuals with lower leg, foot, and ankle musculoskeletal disorders. Thus instrument included 2 subscales: 1) Activities of Daily Living (ADLs) with 21 items and 2) Sports with 8 items. For each subscale patients are asked to answer each question with a single response that most clearly describes their condition within past week. To calculate the score for either subscale, the total number of points are added, divided by the total number os possible points (ADLs-84; Sports-32) and then multiplied by 100.
Hip Disability and Osteoarthritis Outcome Score | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the hip disability and osteoarthritis outcome score (HOOS) Scoring Formula: 100 - [(patient's score of the subscale x 100)/(total score of the subscale)]
Knee Injury and Osteoarthritis Outcome Score | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in condition-specific clinical outcomes over time measured through the Knee Injury and Osteoarthritis Outcome Score (KOOS) Scoring Formula: 100 - [(patient's score of the subscale x 100)/(total score of the subscale)]

SECONDARY OUTCOMES:
Self-reported Pain | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Pain Numerical Rating Scale
Self-reported Surgical Intent | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through a 0-10 Surgical Intent Numerical Rating Scale
Self-reported Medication | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through self reported consumption of painkillers
Anxiety | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through the General Anxiety Disorder-7 (GAD7) scale.
Depression | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Self-administered version of the PRIME-MD diagnostic instrument for common mental disorders, used to monitor the severity of depression and response to treatment. The PHQ-9 is the depression module, which scores each of the nine DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Validated for use in primary care.
Fear avoidance behaviour | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through the Fear Avoidance Beliefs Questionnaire - Work & Physical Activity (FABQ).
Work Productivity and Absenteeism | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change over time in clinical outcomes common to all conditions measured through the Work Productivity and Activity Impairment Questionnaire (WPAI).
Engagement levels | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in patient interaction with medical device over time measured through adherence levels. Patients are asked to perform daily therapeutic sessions, 5-7 days a week. Engagement is calculated weekly and averaged by the end of the therapeutic program.
Satisfaction scores | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in patient interaction with medical device over time measured through Net Promoter Scores. Patients are asked to report their satisfaction level by answering the question: "On a scale from zero to ten, how much would you recommend the system to one of your friends or neighbours?", where 0=do not recommend at all and 10=highly recommend.
Completion rates | Baseline, each four weeks after initiation of rehabilitation program, and periodical follow-up assessments (each 8 weeks) until 2 years after enrolment
  Change in patient interaction with medical device over time measured through average retention rates at 8/12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando D Correia, MD, Principal Investigator — Centro Hospitalar e Universitário do Porto
Locations (1):
- SWORD Health Technologies, Inc, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and study aggregate results (including anonymised individual patient data) will be made available
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available upon study publication, for 5 years.
Access Criteria: Study protocol will be available through a direct link in this platform. The excel file with the aggregate results will be made available as supplementary information upon study publication.

REFERENCES:
- [Derived] C Areias A, G Moulder R, Molinos M, Janela D, Bento V, Moreira C, Yanamadala V, P Cohen S, Dias Correia F, Costa F. Predicting Pain Response to a Remote Musculoskeletal Care Program for Low Back Pain Management: Development of a Prediction Tool. JMIR Med Inform. 2024 Nov 19;12:e64806. doi: 10.2196/64806. PMID 39561359
- [Derived] Areias AC, Janela D, Molinos M, Bento V, Moreira C, Yanamadala V, Cohen SP, Correia FD, Costa F. Exploring the Importance of Race and Gender Concordance Between Patients and Physical Therapists in Digital Rehabilitation for Musculoskeletal Conditions: Observational, Longitudinal Study. J Med Internet Res. 2024 Oct 29;26:e65354. doi: 10.2196/65354. PMID 39470695
- [Derived] Janela D, Areias AC, Moulder RG, Molinos M, Bento V, Yanamadala V, Correia FD, Costa F. Recovering Work Productivity in a Population With Chronic Musculoskeletal Pain: Unveiling the Value and Cost-Savings of a Digital Care Program. J Occup Environ Med. 2024 Oct 1;66(10):e493-e499. doi: 10.1097/JOM.0000000000003191. Epub 2024 Jul 16. PMID 39016261
- [Derived] Scheer J, Areias AC, Molinos M, Janela D, Moulder R, Lains J, Bento V, Yanamadala V, Dias Correia F, Costa F. Engagement and Utilization of a Complete Remote Digital Care Program for Musculoskeletal Pain Management in Urban and Rural Areas Across the United States: Longitudinal Cohort Study. JMIR Mhealth Uhealth. 2023 Mar 16;11:e44316. doi: 10.2196/44316. PMID 36735933
- [Derived] Areias AC, Costa F, Janela D, Molinos M, Moulder RG, Lains J, Scheer JK, Bento V, Yanamadala V, Cohen SP, Correia FD. Impact on productivity impairment of a digital care program for chronic low back pain: A prospective longitudinal cohort study. Musculoskelet Sci Pract. 2023 Feb;63:102709. doi: 10.1016/j.msksp.2022.102709. Epub 2022 Dec 12. PMID 36543719
- [Derived] Janela D, Costa F, Molinos M, Moulder RG, Lains J, Bento V, Scheer JK, Yanamadala V, Cohen SP, Correia FD. Digital Rehabilitation for Elbow Pain Musculoskeletal Conditions: A Prospective Longitudinal Cohort Study. Int J Environ Res Public Health. 2022 Jul 27;19(15):9198. doi: 10.3390/ijerph19159198. PMID 35954555
- [Derived] Costa F, Janela D, Molinos M, Moulder R, Bento V, Lains J, Scheer J, Yanamadala V, Cohen S, Dias Correia F. Impacts of Digital Care Programs for Musculoskeletal Conditions on Depression and Work Productivity: Longitudinal Cohort Study. J Med Internet Res. 2022 Jul 25;24(7):e38942. doi: 10.2196/38942. PMID 35714099
- [Derived] Costa F, Janela D, Molinos M, Lains J, Francisco GE, Bento V, Dias Correia F. Telerehabilitation of acute musculoskeletal multi-disorders: prospective, single-arm, interventional study. BMC Musculoskelet Disord. 2022 Jan 4;23(1):29. doi: 10.1186/s12891-021-04891-5. PMID 34983488